CLINICAL TRIAL: NCT01581905
Title: A Randomized Controlled Trial Comparing Conventional Laparoscopic Hysterectomy With Robot-Assisted Laparoscopic Hysterectomy at a Teaching Institution
Brief Title: Study of Conventional Laparoscopic Hysterectomy Versus Robot-Assisted Laparoscopic Hysterectomy at a Teaching Institution
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was redesigned as a new trial
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38824
Record Dates: First submitted 2012-02-24; First posted 2012-04-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Menorrhagia; Dysfunctional Uterine Bleeding; Leiomyoma; Pelvic Pain; Endometriosis
Keywords: Hysterectomy; Laparoscopy; Robotics
MeSH Terms: conditions — Menorrhagia; Metrorrhagia; Leiomyoma; Pelvic Pain; Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LH Group (Active Comparator): The LH Group includes individuals undergoing conventional laparoscopic hysterectomy, total or supracervical.
  Interventions: Procedure: Conventional Laparoscopic Hysterectomy (LH)
- RH Group (Active Comparator): The RH Group includes individuals undergoing Robot-Assisted laparoscopic hysterectomy, total or supracervical.
  Interventions: Procedure: Robot Assisted Hysterectomy

INTERVENTIONS:
Procedure: Conventional Laparoscopic Hysterectomy (LH) — Patients assigned to this intervention will undergo conventional laparoscopic hysterectomy, either total or supracervical.
  Other Names: LH Group
  Arms: LH Group
Procedure: Robot Assisted Hysterectomy — Patients assigned to this group will undergo Robot-Assisted Laparoscopic Hysterectomy, either total or supracervical.
  Other Names: RH Group
  Arms: RH Group

SUMMARY:
Approximately 600,000 women undergo hysterectomy each year in the United States, of which 12% are laparoscopic. The most common indications for hysterectomy are: symptomatic uterine leiomyomas (40.7%), endometriosis (17.7%), and prolapse (14.5%). The first total laparoscopic hysterectomy was performed by Reich et al in 1988. Many studies have proven that laparoscopic hysterectomy is associated with lower preoperative morbidity, shorter hospital stay, and shorter recovery times than abdominal hysterectomy. The literature has also shown the complication rates for laparoscopic cases are similar to open procedures in the hands of an experienced laparoscopic surgeon. The American Congress of Obstetricians and Gynecologists Committee on Gynecologic Practice state that laparoscopic hysterectomy is an alternative to abdominal hysterectomy for those patients in whom vaginal hysterectomy is not indicated or feasible. The ACOG Committee on Gynecologic Practice site multiple advantages of laparoscopic hysterectomy to abdominal hysterectomy including faster recovery, shorter hospital stay, less blood loss, and fewer abdominal wall/wound infections. Despite the recommendations of ACOG for a more minimally invasive approach, 66% of all hysterectomies are performed abdominally. Key reasons for the lag in utilization of laparoscopic techniques are the technical obstacles of performing minimally invasive hysterectomies. Robotic technology has emerged as a means to decrease the learning curve and increase the availability of minimally invasive surgery to patients. A current review of the literature reveals no randomized trials evaluating the efficacy of conventional laparoscopic hysterectomy vs. robot-assisted laparoscopic hysterectomy. The investigator's aim is to address this void.

The primary objective of this study is to determine whether Robot-Assisted Laparoscopic Hysterectomy is equivalent to Conventional Laparoscopic Hysterectomy with respect to operative time, blood loss, and hospital stay. The investigator's secondary objective was to assess the cost, morbidity, and mortality of each procedure.

DETAILED DESCRIPTION:
See Above

ELIGIBILITY:
Inclusion Criteria:

* Individuals recruited into this study will be patients presenting to the Urogynecology and Minimally Invasive Surgical Group for consultation for hysterectomy.

Exclusion Criteria:Individuals who are not candidates for laparoscopic surgery

* Medical Condition that does not allow pneumoperitoneum
* Medical Condition that does not allow proper ventilation during anesthesia
* Uterine size precluding access to the uterine artery
* Pelvic Organ Prolapse amendable to a vaginal approach

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Operating Time | Operating time is measured on the day of surgery after completing the procedure.

SECONDARY OUTCOMES:
Estimated Blood Loss | Estimated blood loss will be measured on the day of surgery after completing the procedure.
Intraoperative Complications | Intraoperative complications will be measured on the day of surgery after completing the procedure.
  Intraoperative complications include: injury to bladder, ureters, bowel, blood vessels,and nerves AND hemorrhage
Perioperative Complications | Perioperative complications will be measured on the date of discharge from the hospital.
  Perioperative complications include: urinary tract infections, urinary retention, ileus, myocardial infarction, atrial fibrillation, pulmonary edema, atelectasis, pneumonia, renal and cerebrovascular morbidity, thromboembolic complications (DVT and PE)
Early Postoperative Complications | Early postoperative complications will be measured on the date of discharge from the hospital until two weeks after surgery, assessed up to 14 days post-operativley.
  Early postoperative complications include: pulmonary, renal, and cerebrovascular morbidity, wound and vault complications (infection, breakdown, and dehiscence); septicemia, and thromboembolic complications (DVT, PE)
Delayed Post-Operative Complications | Delayed post-operative complications will be measured from 2 weeks until 8 weeks after surgery, up to 56 days post-operatively.
  Delayed post-operative complications include: incisional hernia formation, re-operation, vaginal evisceration
Costs | Cost will be assessed 8 weeks after completion of the surgery, up to 56 days post-operatively.
  Costs will include the costs of pre-operative care, surgery, post-operative care, and any post-operative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Janis L Green, MD, Principal Investigator — Milton S. Hershey Medical Center; Gerald J Harkins, MD, Study Director — Milton S. Hershey Medical Center; Matthew Davies, MD, Study Chair — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Sarlos D, Kots LA. Robotic versus laparoscopic hysterectomy: a review of recent comparative studies. Curr Opin Obstet Gynecol. 2011 Aug;23(4):283-8. doi: 10.1097/GCO.0b013e328348a26e. PMID 21666467
- [Background] Pasic RP, Rizzo JA, Fang H, Ross S, Moore M, Gunnarsson C. Comparing robot-assisted with conventional laparoscopic hysterectomy: impact on cost and clinical outcomes. J Minim Invasive Gynecol. 2010 Nov-Dec;17(6):730-8. doi: 10.1016/j.jmig.2010.06.009. Epub 2010 Sep 17. PMID 20850391
- [Background] Payne TN, Dauterive FR. A comparison of total laparoscopic hysterectomy to robotically assisted hysterectomy: surgical outcomes in a community practice. J Minim Invasive Gynecol. 2008 May-Jun;15(3):286-91. doi: 10.1016/j.jmig.2008.01.008. Epub 2008 Mar 6. PMID 18439499
- [Background] Sarlos D, Kots L, Stevanovic N, Schaer G. Robotic hysterectomy versus conventional laparoscopic hysterectomy: outcome and cost analyses of a matched case-control study. Eur J Obstet Gynecol Reprod Biol. 2010 May;150(1):92-6. doi: 10.1016/j.ejogrb.2010.02.012. Epub 2010 Mar 5. PMID 20207063
- [Background] Shashoua AR, Gill D, Locher SR. Robotic-assisted total laparoscopic hysterectomy versus conventional total laparoscopic hysterectomy. JSLS. 2009 Jul-Sep;13(3):364-9. PMID 19793478